CLINICAL TRIAL: NCT04076436
Title: Efficacy of Intravenous Fosfomycin in the Treatment of Complicated Urinary in Real-life Conditions. Impact of the CMI and Baseline Mutations. FOSFO-MIC Project
Brief Title: Efficacy of Intravenous Fosfomycin in the Treatment of Complicated Urinary in Real-life Conditions.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-FOS-2019-01
Record Dates: First submitted 2019-08-22; First posted 2019-09-03 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-08

CONDITIONS: Complicated Urinary Tract Infection
Keywords: Prospective follow-up study; Real-life conditions; Complicated urinary tract infection; Escherichia coli infection; Fosfomycin efficacy; Quinolones; Beta-lactams; Microbiological failure; Resistance development
MeSH Terms: conditions — Escherichia coli Infections | interventions — beta-Lactams

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fosfomycin cohort:: Cohort of patients with complicated urinary tract infection caused by Escherichia coli treated with intravenous fosfomycin
  Interventions: Other: Drug: Intravenous fosfomycin
- Quinolones or beta-lactams cohort: Cohort of patients with complicated urinary tract infection caused by Escherichia coli treated with intravenous quinolones or beta-lactams.
  Interventions: Other: Drug: Intravenous quinolone or beta-lactam

INTERVENTIONS:
Other: Drug: Intravenous fosfomycin — Patients will be visited on days 1 (Day of the urine and blood culture taking), 2, 5, 7, 14, on the test of cure and on day 30.
  Visit on day 1: First day of treatment. Basal data collection.
  Visit on day 2: Blood collection to fosfomycin levels calculation.
  Visits on days 5, 7, 14, on the test of cure (day 21): Clinical evolution data, Urocultures and Adverse effects.
  Visit on day 30: Assess mortality
  Groups: Fosfomycin cohort:
Other: Drug: Intravenous quinolone or beta-lactam — Patients will be visited on days 1 (Day of the urine and blood culture taking), 5, 7, 14, on the test of cure and on day 30.
  Visit on day 1: First day of treatment. Basal data collection.
  Visits on days 5, 7, 14, on the test of cure (day 21): Clinical evolution data, Urocultures and Adverse effects.
  Visit on day 30: Assess mortality
  Groups: Quinolones or beta-lactams cohort

SUMMARY:
This will be a prospective observational multicentre study in real-life conditions of patients with complicated urinary infection of community presentation caused by Escherichia coli using intravenous fosfomycin, quinolones or beta-lactams.

It's a multicenter and multinational study and it will include 200 patients in the fosfomycin cohort and 200 patients in the control cohort (quinolones or beta-lactams).

DETAILED DESCRIPTION:
The objectives are:

1. To asses the clinical and microbiological efficacy and safety of intravenous fosfomycin in the treatment of complicated urinary tract infections due to Escherichia coli in real life conditions, in comparison with a matched cohort of patients treated with quinolones or beta-lactams.
2. To evaluate the frequency of microbiological failure and development of resistance (or decrease in sensitivity) in Escherichia coli isolates, depending on different pharmacokinetic and pharmacodynamic parameters, with special emphasis on fAUC0-24/MIC.
3. To evaluate the frequency of microbiological failure and development of resistance (or decrease in sensitivity) and their association with the existence of basal mutations in genes related to intracellular transport or regulation of these transporters.

For objective 1, a study of prospective mated cohorts (fosfomycin cohort versus quinolones or beta-lactams cohort) will be performed, and for objectives 2 and 3 a prospective cohort study (fosfomycin cohort) will be conducted.

ELIGIBILITY:
Fosfomycin cohort:

* Inclusion criteria: Patients over 18 years of age. Patients who have started treatment with intravenous fosfomycin, estimated that they will require at least 2 days of treatment with fosfomycin, initiated as either as empirical treatment (within 24 hours after the emergency visit or onset of symptoms) or targeted treatment (within 24 hours of the availability of the antibiogram).
* Exclusion criteria: Patients under 18 years of age. Patients in palliative treatment.

Control cohort (objective 1):

* Inclusion criteria:Patients over 18 years of age. Patients who have started treatment with intravenous quinolones or beta-lactams, estimated that they will require at least 2 days of treatment with the drug, initiated as either as empirical treatment (within 24 hours after the emergency visit or onset of symptoms) or targeted treatment (within 24 hours of the availability of the antibiogram). Each patient from the fosfomycin cohort will be matched with a patient from this control cohort according to their.
* Exclusion criteria: Patients under 18 years of age.Patients in palliative treatment; Informed consent not signed by the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with complicated urinary tract infection
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-10-21 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference in the proportion of subjects getting clinical-microbiological cure on the test of cure between the fosfomycin cohort and the quinolones or beta-lactams cohort | 21 days
  The difference in the proportion of subjects getting clinical-microbiological cure (disappearance of all new symptoms or signs related to urinary infection and negative uroculture) on the test of cure between the fosfomycin cohort and the quinolones or beta-lactams cohort
The proportion of microbiological failure on the test of cure in the fosfomycin cohort (measured as isolation of Escherichia coli in uroculture on the test of cure). | 21 days
  The proportion of microbiological failure on the test of cure in the fosfomycin cohort (measured as isolation of Escherichia coli in uroculture on the test of cure).
The proportion of development of resistance (or decrease in sensitivity) to fosfomycin during or after treatment: Presence of mutation in genes uhpT, uhpA, uhpB, uhpC, uhpT, crp, cyaA, ptsl and fosA and measure CMI. | 30 days
  The proportion of development of resistance (or decrease in sensitivity) to fosfomycin during or after treatment: Presence of mutation in genes uhpT, uhpA, uhpB, uhpC, uhpT, crp, cyaA, ptsl and fosA and measure CMI.

SECONDARY OUTCOMES:
To evaluate the frequency of microbiological failure and development of resistance (or decrease in sensitivity) in Escherichia coli isolates. | 30 days
  To evaluate the frequency of microbiological failure and development of resistance (or decrease in sensitivity) in Escherichia coli isolates.
The difference in the proportion of solicited EAs in subjects in fosfomycin cohort and quinolones or beta-lactams cohort. | Day 5 through Day 21
  The difference in the proportion of solicited EAs in subjects in fosfomycin cohort and quinolones or beta-lactams cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Belén Gutiérrez Gutiérrez, Study Director — Hospital Universitario Virgen Macarena
Locations (2):
- Spain (2):
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario Virgen Macarena, Seville